CLINICAL TRIAL: NCT00434954
Title: Effect of Exenatide Plus Metformin vs. Premixed Human Insulin Aspart Plus Metformin on Glycemic Control and Hypoglycemia in Patients With Inadequate Control of Type 2 Diabetes on Oral Antidiabetic Treatment
Brief Title: Effect of Exenatide Plus Metformin vs. Insulin Aspart Plus Metformin on Glycemic Control and Hypoglycemia in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-SB-GWBN
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Results first posted 2010-08-23 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — BID protein, human; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide Twice Daily (BID) (Experimental)
  Interventions: Drug: exenatide twice daily (BID)
- Premixed Insulin Aspart Twice Daily (BID) (Active Comparator)
  Interventions: Drug: premixed insulin aspart twice daily (BID)

INTERVENTIONS:
Drug: exenatide twice daily (BID) — subcutaneous injection (5 mcg or 10 mcg), twice a day
  Other Names: Byetta
  Arms: Exenatide Twice Daily (BID)
Drug: premixed insulin aspart twice daily (BID) — subcutaneous injection (titrated appropriately), twice a day
  Arms: Premixed Insulin Aspart Twice Daily (BID)

SUMMARY:
This study in Germany is designed to compare the effects of twice-daily exenatide plus metformin and twice-daily premixed human insulin aspart plus metformin with respect to glycemic control, as measured by HbA1c, combined with the percentage of patients with at least one treatment-emergent hypoglycemic episode. Patients will be treated with study therapy for approximately 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have been treated with diet and exercise and a stable, maximally tolerated dose of immediate-release or extended-release metformin, or the combination of metformin (any dosage) with sulfonylurea/meglitinides for at least 3 months prior to study start
* Have not received thiazolidinediones, or alpha-glucosidase inhibitors for longer than 2 weeks within 3 months prior to study start, and have not received any insulin formulation for more than 14 days (other than in emergency situations) and within 14 days prior to study start
* Have an HbA1c between 6.5% and 10.0%, inclusive
* Have a body mass index (BMI) between 25 kg/m^2 and 40 kg/m^2, inclusive

Exclusion Criteria:

* Have type 1 diabetes or known latent autoimmune diabetes in adults
* Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks prior to study start
* Are receiving treatment for gastrointestinal disease with a drug directly affecting gastrointestinal motility (e.g., metoclopramide, cisapride, and chronic macrolide antibiotics)
* Have used any prescription drug to promote weight loss within 3 months prior to study start
* Have received treatment within 30 days prior to study start with a drug that has not received regulatory approval for any indication at the time of study entry
* Have previously completed or withdrawn from this study or any other study investigating exenatide or GLP-1 analogs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (39):
- Germany (39):
  - Research Site, Bad Mergentheim
  - Research Site, Berlin
  - Research Site, Bosenheim
  - Research Site, Burghausen
  - Research Site, Datteln
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Friedrichsthal
  - Research Site, Hildesheim
  - Research Site, Hirschhorn
  - Research Site, Hohenmölsen
  - Research Site, Jena
  - Research Site, Lehrte
  - Research Site, Leipzig
  - Research Site, Ludwigsburg
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, Marktheidenfeld
  - Research Site, Meissen
  - Research Site, München
  - Research Site, Offenbach
  - Research Site, Oschatz
  - Research Site, Pohlheim
  - Research Site, Regensburg
  - Research Site, Riesa
  - Research Site, Rodgau
  - Research Site, Roding
  - Research Site, Rosenheim
  - Research Site, Schlüchtern
  - Research Site, Schwedt
  - Research Site, Sinsheim
  - Research Site, Speyer
  - Research Site, Unterhaching
  - Research Site, Völklingen
  - Research Site, Wallerfing
  - Research Site, Wangen
  - Research Site, Warburg
  - Research Site, Wiesbaden
  - Research Site, Wolfsburg

REFERENCES:
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- [Derived] Gallwitz B, Bohmer M, Segiet T, Molle A, Milek K, Becker B, Helsberg K, Petto H, Peters N, Bachmann O. Exenatide twice daily versus premixed insulin aspart 70/30 in metformin-treated patients with type 2 diabetes: a randomized 26-week study on glycemic control and hypoglycemia. Diabetes Care. 2011 Mar;34(3):604-6. doi: 10.2337/dc10-1900. Epub 2011 Feb 1. PMID 21285388

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients treated with metformin (MET only;confirmatory population used for primary analysis) and additional patients treated with metformin plus either sulfonylurea or meglitinide (MET+SU; exploratory population) were enrolled at a 3:1 ratio; metformin was continued.Within each population, patients were then randomly assigned 1:1 to study treatment
Groups:
- Exenatide Twice Daily: Exenatide 5 mcg twice daily for 4 weeks, followed by 10 mcg twice daily for 26 weeks
- Premixed Insulin Aspart Twice Daily: Premixed insulin aspart (70% protamin crystallized, 30% soluble) twice daily, individually titrated to reach target blood glucose levels for 26 weeks
Period: Overall Study
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Started | 248 | 246
Started - Previous Treatment MET Only | 182 | 181
Started - Previous Treatment MET + SU | 66 | 65
Full Analysis Set (FAS) Overall | 247 (FAS=received >=1 dose of study drug. Adverse event data reported for Overall FAS.) | 233 (FAS=received >=1 dose of study drug. Adverse event data reported for Overall FAS.)
FAS - Previous Treatment MET Only | 181 (Baseline and efficacy data reported for "FAS-Previous Treatment MET Only" group.) | 173 (Baseline and efficacy data reported for "FAS-Previous Treatment MET Only" group.)
FAS - Previous Treatment MET + SU | 66 | 60
Completed - Previous Treatment MET Only | 135 | 137
Completed - Previous Treatment MET + SU | 31 | 38
Completed | 166 | 175
Not Completed | 82 | 71
Not completed — Adverse Event | 17 | 2
Not completed — Entry criteria not met | 14 | 16
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 6 | 3
Not completed — Protocol Violation | 36 | 27
Not completed — Sponsor decision | 1 | 0
Not completed — Subject decision | 8 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily | Total
Number analyzed (Participants) | 181 | 173 | 354
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 138 | 133 | 271
  >=65 years | 43 | 40 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.03) | 56.9 (9.94) | 57.1 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 77 | 150
  Male | 108 | 96 | 204
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg / m^2] | 33.4 (4.23) | 32.9 (4.37) | 33.2 (4.30)
Body Weight [Mean (Standard Deviation); unit: kg] | 99.4 (16.22) | 96.6 (17.40) | 98.0 (16.85)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 4.8 (4.39) | 5.2 (4.67) | 5.0 (4.53)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage] | 7.89 (0.822) | 7.88 (0.918) | 7.88 (0.869)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Change in HbA1c from baseline after 26 weeks of treatment (i.e., HbA1c at week 26 minus HbA1c at week 0)
Time Frame: Baseline and 26 weeks
Population: All randomized patients who were previously treated with metformin only and who received at least one dose of study drug (MET only, FAS) and had baseline and at least one post-baseline value available
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
Percentage of glycosylated hemoglobin | -1.00 (0.05) | -1.14 (0.05)
Statistical Analysis 1: Comparison: Exenatide Twice Daily vs Premixed Insulin Aspart Twice Daily; The hypothesis was tested hierarchically that 1) exenatide BID is non-inferior to insulin aspart 70/30 BID for glycemic control (change in HbA1c, outcome measure 1), and 2) superior regarding the incidence of hypoglycemia (outcome measure 2). This is the first part of the hierarchical test; Test type: Non-Inferiority or Equivalence — The planned sample size of 366 patients treated with metformin only (assuming 25% dropouts) gave a power of 85% to detect non-inferiority of exenatide BID for change in HbA1c (non-inferiority margin 0.4%; assumed common standard deviation of 1.1%); p = 0.055, Mixed effect model repeat measures(MMRM) — Non-inferiority: upper limit of 95% Confidence Interval (CI) to be < 0.4%; 95% CI of treatment group difference derived from MMRM (treatment, week, baseline HbA1c and interactions as fixed effects); p-value: superiority test; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.003 to 0.291]

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of < 6.5%
Description: Percentage of subjects achieving HbA1c target of < 6.5% at the end of study (week 26) [i.e., number of subjects who achieved HbA1c < 6.5% divided by total number of subjects times 100%].
Time Frame: 26 weeks
Population: All randomized patients who were previously treated with metformin only and who received at least one dose of study drug (MET only, FAS); last observation carried forward
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
Percentage of participants | 27.6 | 24.9
Statistical Analysis 1: Comparison: Exenatide Twice Daily vs Premixed Insulin Aspart Twice Daily; Test type: Superiority or Other; p = 0.554, Chi square test (Pearson)

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of < 7.0%
Description: Percentage of subjects achieving HbA1c target of < 7.0% at the end of study (week 26) [i.e., number of subjects who achieved HbA1c < 7.0% divided by total number of subjects times 100%].
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
Percentage of participants | 49.2 | 56.6
Statistical Analysis 1: Comparison: Exenatide Twice Daily vs Premixed Insulin Aspart Twice Daily; Test type: Superiority or Other; p = 0.159, Chi square test (Pearson)

4. Secondary Outcome: Incidence of Hypoglycemic Episodes [Blood Glucose <= 3.0 mmol/L or Severe] (Percentage of Subjects Who Experienced at Least One Treatment-emergent Hypoglycemic Episode During the 26-week Treatment Period)
Description: Risk for the first hypoglycemic episode to occur up to Week 26 (percentage of subjects who experienced at least one treatment-emergent hypoglycemic episode during the 26-week treatment period)[ i.e., number of subjects experiencing at least one hypoglycemic episode divided by total number of subjects times 100%]
Time Frame: 26 weeks
Population: All randomized patients who were previously treated with metformin only and who received at least one dose of study drug (MET only, FAS)
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
Percentage of participants | 1.8 | 6.3

5. Secondary Outcome: Incidence of Nocturnal Hypoglycemia (Percentage of Subjects Who Experienced at Least One Episode of Nocturnal Hypoglycemia During the 26 Week Treatment Period)
Description: Risk for first nocturnal (night-time) hypoglycemic episode to occur up to week 26 (percentage of subjects who experienced at least one episode of nocturnal hypoglycemia during the 26 week treatment period) [i.e., number of subjects who experienced nocturnal hypoglycemia divided by total number of subjects times 100%].
Time Frame: 26 weeks
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
Percentage of participants | 3.9 | 7.0

6. Secondary Outcome: 7 Point Self-monitored Blood Glucose (SMBG) Profiles
Description: 7-point self-monitored blood glucose profiles at baseline and the end of the study, measured at 7 times during the day (pre-breakfast, 2 hours post-breakfast, pre-lunch, 2 hours post-lunch, pre-dinner, 2 hours post-dinner, and 3:00am).
Time Frame: Baseline and 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
mg/dL
  Pre-breakfast at baseline (week 0) | 8.933 (1.7138) | 9.005 (2.0432)
  Pre-breakfast at endpoint (week 26) | 7.774 (1.7730) | 7.293 (1.3349)
  2 hrs post-breakfast at baseline (week 0) | 10.821 (2.5306) | 10.902 (2.8499)
  2 hrs post-breakfast at endpoint (week 26) | 8.014 (2.0557) | 8.304 (2.1212)
  Pre-lunch at baseline (week 0) | 8.443 (2.1814) | 8.357 (2.3221)
  Pre-lunch at endpoint (week 26) | 7.506 (1.8800) | 6.656 (1.7011)
  2 hrs post-lunch at baseline (week 0) | 9.698 (2.2370) | 9.899 (2.6433)
  2 hrs post-lunch at endpoint (week 26) | 8.513 (5.8997) | 8.216 (1.6108)
  Pre-dinner at baseline (week 0) | 8.684 (2.0059) | 8.759 (2.2174)
  Pre-dinner at endpoint (week 26) | 7.616 (2.1727) | 7.194 (1.5572)
  2 hrs post-dinner at baseline (week 0) | 10.241 (2.2880) | 10.259 (2.4868)
  2 hrs post-dinner at endpoint (week 26) | 7.727 (1.8820) | 8.143 (1.5614)
  3:00 am at baseline (week 0) | 8.323 (1.8692) | 8.475 (2.2643)
  3:00 am at endpoint (week 26) | 7.518 (1.5861) | 6.999 (1.5596)

7. Secondary Outcome: Blood Lipid Levels
Description: Total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol (calculated), and triglyceride levels at baseline (week 0) and the end of the study (week 26)
Time Frame: Baseline and 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
mmol/L
  Total cholesterol at baseline (week 0) | 5.147 (1.0008) | 5.084 (1.0079)
  Total cholesterol at endpoint (week 26) | 4.971 (0.9653) | 5.050 (0.8933)
  HDL cholesterol at baseline (week 0) | 1.234 (0.3065) | 1.255 (0.3324)
  HDL cholesterol at endpoint (week 26) | 1.244 (0.2805) | 1.319 (0.3394)
  LDL cholesterol (calculated) at baseline (week 0) | 2.845 (0.8308) | 2.768 (0.8103)
  LDL cholesterol (calculated) at endpoint (week 26) | 2.738 (0.8472) | 2.852 (0.8134)
  Triglycerides at baseline (week 0) | 2.391 (1.5497) | 2.410 (1.4398)
  Triglycerides at endpoint (week 26) | 2.234 (1.1886) | 2.006 (1.2040)

8. Primary Outcome: Incidence of Hypoglycemia (Percentage of Participants With at Least One Hypoglycemic Episode)
Description: Risk for first hypoglycemic episode (blood glucose <=3.9 mmol/L or severe episode) to occur up to week 26
Time Frame: 26 weeks
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
Percentage of participants | 8.0 | 20.5
Statistical Analysis 1: Comparison: Exenatide Twice Daily vs Premixed Insulin Aspart Twice Daily; The hypothesis was tested hierarchically that 1) exenatide BID is non-inferior to insulin aspart BID for glycemic control (outcome measure 1), and 2) superior regarding the incidence of hypoglycemia (outcome measure 2).The planned sample size of 366 patients treated with metformin only (assumed dropout rate 25%) gave 96% power to detect superiority of exenatide BID for the risk of hypoglycemia, assuming incidences of 3.6% for exenatide BID and 17.5% for insulin aspart BID (alpha=0.05); Test type: Superiority or Other; p < 0.05, Kaplan-Meier analysis — Non overlapping 95% CI's: statistically significant difference p<0.05; For each treatment group, the incidence of hypoglycemia at Week 26 and 95% CIs were derived from Kaplan-Meier analysis

9. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline after 26 weeks of treatment (i.e., body weight at week 26 minus body weight at week 0)
Time Frame: Baseline and 26 weeks
Population: All randomized patients who were previously treated with metformin only and who received at least one dose of study drug (MET only, FAS) and had baseline and at least one post-baseline value available; last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
kg | -4.10 (0.22) | 1.02 (0.22)
Statistical Analysis 1: Comparison: Exenatide Twice Daily vs Premixed Insulin Aspart Twice Daily; Test type: Superiority or Other; p < 0.0001, Mixed effects model repeated measures — The MMRM model adjusted for baseline HbA1c stratum (HbA1c at baseline >= 6.5% and <= 8.0% vs. > 8.0% and <=10%); 95% CI of treatment group difference derived from MMRM (treatment, week, baseline HbA1c and interactions as fixed effects)

10. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI from baseline after 26 weeks of treatment (i.e., BMI at week 26 minus BMI at week 0)
Time Frame: Baseline and 26 weeks
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
kg/m^2 | -1.39 (0.07) | 0.32 (0.07)
Statistical Analysis 1: Comparison: Exenatide Twice Daily vs Premixed Insulin Aspart Twice Daily; Test type: Superiority or Other; p < 0.0001, Mixed effects model repeated measures — The MMRM model adjusted for baseline HbA1c stratum (HbA1c at Visit 1 >= 6.5% and <= 8.0% vs. > 8.0% and <=10%); [statistical method as in outcome 9, analysis 1]

11. Secondary Outcome: Patient Reported Outcomes: Diabetes Treatment Satisfaction Questionnaire (DTSQ)
Description: Total DTSQ treatment satisfaction score at baseline (week 0) and after 26 weeks of treatment (LOCF). Total DTSQ treatment satisfaction score is derived as sum score of the individual components 1 and 4-8 of the DTSQ questionnaire. Each component is scored on a scale of 0 (worst case) to 6 (best case). Higher values represent higher treatment satisfaction.
Time Frame: Baseline and 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on DTSQ scale
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
scores on DTSQ scale
  DTSQ score at baseline (week 0) | 29.5 (6.13) | 29.7 (6.25)
  DTSQ score at endpoint (week 26) | 30.6 (6.05) | 29.3 (6.59)

12. Secondary Outcome: Patient Reported Outcomes: Quality of Life (SF-12)
Description: SF-12 Physical and Mental Component Summary Scores at baseline (week 0) and after 26 weeks of treatment (LOCF). SF-12 Physical and Mental Component Summary Scores are normalized scores ranging from 0 (worst case) to 100 (best case), and are derived from responses to 12 questions. Scores > 50 indicate an above-average health status.
Time Frame: Baseline and 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on SF-12 scale
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Number analyzed (Participants) | 181 | 173
scores on SF-12 scale
  Physical Component at baseline (week 0) | 35.5 (13.99) | 36.3 (14.45)
  Physical Component at endpoint (week 26) | 39.1 (14.30) | 37.7 (14.28)
  Mental Component at baseline (week 0) | 31.3 (18.33) | 28.3 (19.43)
  Mental Component at endpoint (week 26) | 31.1 (19.38) | 29.6 (18.36)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Exenatide Twice Daily | Premixed Insulin Aspart Twice Daily
Serious Adverse Events (participants affected / at risk) | 9/247 | 8/233
Other Adverse Events (participants affected / at risk) | 102/247 | 66/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Twice Daily (N=247) | Premixed Insulin Aspart Twice Daily (N=233)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Twice Daily (N=247) | Premixed Insulin Aspart Twice Daily (N=233)
Diarrhea (Gastrointestinal disorders) | 27 | 16
Headache (Nervous system disorders) | 26 | 25
Nasopharyngitis (Infections and infestations) | 37 | 42
Nausea (Gastrointestinal disorders) | 46 | 8
Vomiting (Gastrointestinal disorders) | 22 | 2
Dyspepsia (Gastrointestinal disorders) | 15 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days